CLINICAL TRIAL: NCT06002581
Title: Clinical Study on the Efficacy and Safety of rTMS Regulating Slow-wave Sleep to Delay the Progression of Parkinson's Disease
Brief Title: Repetitive Transcranial Magnetic Stimulation(rTMS) Regulating Slow-wave to Delay the Progression of Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xiaoying Zhu, associate chief physician of neurology, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCTR-2022B05
Record Dates: First submitted 2023-07-11; First posted 2023-08-21 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; slow-wave sleep; rTMS; motor symptom; progression
MeSH Terms: conditions — Parkinson Disease; Disease Progression

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the early treatment group (Experimental): stage1+stage2 real stimulation
  Interventions: Device: rTMS real stimulation stage1; Device: rTMS real stimulation stage 2
- the control group (delayed treatment group) (Other): stage1 sham stimulation + stage2 real stimulation
  Interventions: Device: rTMS shame stimulation stage1; Device: rTMS real stimulation stage 2

INTERVENTIONS:
Device: rTMS real stimulation stage1 — In the first stage, the early treatment group use low-frequency rTMS real stimulation,
  Arms: the early treatment group
Device: rTMS shame stimulation stage1 — In the first stage, the control group (delayed treatment group) all use sham stimulation.
  Arms: the control group (delayed treatment group)
Device: rTMS real stimulation stage 2 — In the second stage, both the early treatment group and the control group (delayed treatment group) will be treated with true stimulation low-frequency rTMS.

SUMMARY:
At present, no drug therapy has been proven to delay the progression of Parkinson's disease (PD). rTMS, as a non-invasive neuromodulation method, can regulate Slow-wave sleep (SWS). SWS is recognized closely related to neurodegeneration. However, there has been no clinical studies on if rTMS could delay the progression of PD by regulating SWS.

The main purpose of this study is to explore the changes of SWS in non-rapid eye movement (NREM) sleep period in PD patients by using rTMS, and the relationship with potential improvements of SWS and motor symptom delay. The study aims to find a potential new treatment strategy to delay the neurodegenerative process in PD patients by modulating SWS by rTMS.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the clinically definite or clinically probable PD according to the MDS 2015 version.
2. Chinese Han population (three generations), age greater than or equal to 50 years old, less than or equal to 80 years old, male or female.
3. Hoehn-Yahr stages 1-4.
4. The dose of levodopa drug therapy was stable three weeks before enrollment and during the follow-up period.
5. Right-handed.
6. The patient signed a written informed consent.

Exclusion Criteria:

1. Any form of Parkinsonism other than primary PD.
2. Those who have received neurosurgical intervention or stereotaxic brain surgery for PD, or have previously received TMS treatment.
3. Cognitive dysfunction (MMSE ≤ 24 points) or those who cannot cooperate with the scale score.
4. Persons with mental disabilities.
5. Pregnant women.
6. There are contraindications for rTMS treatment.
7. There are contraindications for MRI examination.
8. Baseline PSG suggests other sleep disorders such as moderate to severe OSAS; BMI>=30.
9. Patients who are addicted to alcohol, taking SSRIs, TCAs, sedative hypnotics, histamine antagonists and other drugs and food that may affect NREM and REM sleep structure.
10. Those who are unwilling to participate in the study or unable to sign the informed consent form; and other circumstances that the researcher considers inappropriate to participate in the study.

    -

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-09-03 (Actual); Primary Completion 2026-07-28 (Estimated); Study Completion 2026-07-28 (Estimated)

PRIMARY OUTCOMES:
Change of Motor Function in PD by Low Frequency rTMS Stimulation | Day14
  the score of Unified Parkinson's Disease Rating ScaleⅢ (UPDRSIII)[off] The higher the score, the more severe the motor dysfunction

SECONDARY OUTCOMES:
Effects of low-frequency rTMS stimulation on motor symptoms | Day28,Day56
  the score of Unified Parkinson's Disease Rating ScaleⅢ (UPDRSIII) [on] The higher the score, the more severe the motor dysfunction
Measurement of improved balance function in patients with Parkinson's disease | Day14,Day28,Day56
  the score of Berg Balance Scale (BBS)[0-56] The higher the score, the better the balance
Assessment of sleep structure in patients with Parkinson's disease | Day14,Day28,Day56
  Use polysomnography (PSG) to record the proportion of slow-wave sleep
Effects of low-frequency rTMS stimulation on anxiety | Day14,Day28,Day56
  the score of Hamilton Anxiety Rating Scale（HAMA)[0-64] The higher the score, the more anxious
Effects of low-frequency rTMS stimulation on cognition | Day14,Day28,Day56
  the score of Montreal Cognitive Assessment（Moca)[0-30] The lower the score, the more severe the cognitive dysfunction
Effects of low-frequency rTMS stimulation on cortical excitability | Day14,Day28
  short-interval cortical inhibition(SICI)
Effects of low-frequency rTMS stimulation on depression | Day14,Day28,Day56
  the score of Hamilton Depression Rating Scale（HAMD） Total score ≥ 20 points: may be mild or moderate depression; The higher the score, the more depressed
Assessment of daytime sleepiness in patients with Parkinson's disease | Day14,Day28,Day56
  the score of The Epworth Sleeping Scale(ESS)[0-24] The higher the score, the more lethargic
Effects of low-frequency rTMS stimulation on gait | Day14,Day28,Day56
  Use a quantitative gait analysis system to analyze the change of gait

OTHER OUTCOMES:
Effects of low-frequency rTMS stimulation on brain connectivity in the PD brain | Day0,Day14,Day28
  functional magnetic resonance imaging (fMRI) (Default mode network, DMN）
Changes in salivary melatonin levels | Day0,Day14,Day28,Day56
  salivary melatonin levels(Fasting)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoying Zhu, doctor, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China